CLINICAL TRIAL: NCT01412125
Title: Study of Biomarkers That Predict the Evolution of Huntington's Disease
Acronym: BIOHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P090302
Record Dates: First submitted 2011-06-23; First posted 2011-08-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Huntington Disease
Keywords: Biomarkers; Genetic polymorphism; Neuroimaging markers; Neuropsychology
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood (for DNA analysis) and plasma sample at inclusion visit
  * Plasma sample every year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patient: Voluntary Huntington patients symptomatic or asymptomatic, with a number of nucleotide expansion(CAG) ≥36 and who know their genetic status
  Interventions: Other: Huntington patient evaluation
- Healthy subject: Voluntary controls with no family history of huntington's disease
  Interventions: Other: Healthy subject evaluation

INTERVENTIONS:
Other: Huntington patient evaluation — Neurological, neuropsychological, neuroimaging evaluation and biological sample
  Groups: Patient
Other: Healthy subject evaluation — Neurological, neuropsychological, neuroimaging evaluation and biological sample
  Groups: Healthy subject

SUMMARY:
Huntington's disease (HD) is a rare, autosomal dominant, progressive neurodegenerative disorder typically becoming noticeable in middle age. It is clinically characterized by progressive involuntary movements (bradykinesia and hyperkinesia), neuropsychiatric disturbances (depression, irritability), and cognitive impairments progressing to dementia.

The striatum (caudate and putamen) is the primary area of neuronal degeneration in HD. Today, there is no validated curative treatment. HD affects approximately 6 000 patients in France and more than 30 000 individuals are considered at risk for this disease.

While the disease gene is discovered and we are capable to do a predictive genetic diagnosis for asymptomatic patients, there is no clinical or biological way to predict the age of onset or the progressive profile of patients.

One of the fundamental characteristics of this disease is its extreme variability from one patient to other both in terms of their evolution and their onset of action. Thus, this inter-individual variability severely limits the genetic counselling and complicating the neurological assessment.

Increasingly, it has been assumed that modifier genes may be the source of this inter-individual variability and that their identification could help the understanding and prediction of disease progression.

Given that the mutant protein is ubiquitous, the molecular dysfunction of neurons could be found in peripheral cells from the bloodstream and will be more accessible to investigation.

DETAILED DESCRIPTION:
In this context, we propose to focus our research not only on biological and genetic markers but also on neuroimaging and neuropsychological markers using paradigms of time reactions or measurement of evoked potentials. We hope to identify sensitive markers of the degenerative process of Huntington's disease even when patients carrying the gene may or may not have reported the disease.

The project is centered on 2 axes:

1. identification of the genetic polymorphism which may explain the phenotypic variability seeing in Huntington's disease
2. identification of biological, genetic and imaging biomarkers that could be used as predictors of clinical progression of Huntington's disease This research is based on the existence of a well followed and well characterized cohort of patients through the Francophone Huntington Network ("RESEAU HUNTINGTON de LANGUE FRANCAISE", RHLF). Therefore, this will help to combine the clinical and biological expertise of RHLF.

ELIGIBILITY:
Inclusion Criteria (patient):

* Voluntary patients symptomatic or asymptomatic
* Patient with a number of CAG ≥36)
* Patient who know his genetic status
* Age greater than 18 years or equal to 18 years
* Patient who provided written informed consent

Exclusion Criteria (patient):

- Deterioration of the protocol preventing the understanding of the protocol

Inclusion Criteria (control):

* Voluntary controls with no family history of huntington's disease
* Control with a number of CAG <36
* Age greater than 18 years or equal to 18 years
* Control who provided written informed consent

Exclusion Criteria (control):

- Deterioration of the protocol preventing the understanding of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from Huntington disease (carrying the gene) versus healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2003-09; Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Unified Huntington Disease Rating Scale (UHDRS) | up to 9 years
  The period of follow-up will achieve at the end of 2020

SECONDARY OUTCOMES:
Mattis Dementia Rating Scale | up to 9 years
  The period of follow-up will achieve at the end of 2020
Trail Making test A et B | up to 9 years
  The period of follow-up will achieve at the end of 2020
Hopkins Verbal Learning Test | up to 9 years
  The period of follow-up will achieve at the end of 2020
Categorical Fluency | up to 9 years
  The period of follow-up will achieve at the end of 2020
Language tests | up to 9 years
  The period of follow-up will achieve at the end of 2020
Social cognition tests | up to 9 years
  The period of follow-up will achieve at the end of 2020
Comportment scale | up to 9 years
  The period of follow-up will achieve at the end of 2020
Neuroimaging | up to 9 years
  The period of follow-up will achieve at the end of 2020
Neuropsychological evaluation | up to 9 years
  The period of follow-up will achieve at the end of 2020
Electrophysiological tests | up to 9 years
  The period of follow-up will achieve at the end of 2020

CONTACTS AND LOCATIONS:
Overall Officials: Bachoud-Lévi Anne-Catherine, PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Henri Mondor, Créteil, France

REFERENCES:
- [Derived] Chenain L, Riad R, Fraisse N, Jubin C, Morgado G, Youssov K, Lunven M, Bachoud-Levi AC. Graph methods to infer spatial disturbances: Application to Huntington's Disease's speech. Cortex. 2024 Jul;176:144-160. doi: 10.1016/j.cortex.2024.04.014. Epub 2024 May 17. PMID 38795650